CLINICAL TRIAL: NCT02834806
Title: BioNIR Ridaforolimus Eluting Coronary Stent System (BioNIR) In Coronary Stenosis Trial
Brief Title: BIONICS Israel Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BioNIR-003
Record Dates: First submitted 2016-07-03; First posted 2016-07-15 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2018-03

CONDITIONS: Stenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BioNIR drug eluting stent system (Experimental): BioNIR Ridaforolimus eluting coronary stent system with modified delivery system
  Interventions: Device: BioNIR Ridaforolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: BioNIR Ridaforolimus Eluting Coronary Stent System — BioNIR Ridaforolimus eluting coronary stent system with modified delivery system

SUMMARY:
This study aims to assess the device success and the safety of Medinol's Drug Eluting Stent - BioNIR - with a modified delivery system. The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:

* A mounted Cobalt Chromium (CoCr) alloy based stent
* A Rapid Exchange (RX) delivery system
* A polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
* Ridaforolimus drug - CAS Registry Number: 572924-54-0 It is indicated for improving coronary luminal diameter in patients with symptomatic heart disease due to lesions in vessels with reference diameters of 2.5 mm to 4.25 mm, including complex lesions.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, open label, clinical trial. Lesions planned to be treated must be declared and recorded at time of enrollment. Planned staged procedures, if necessary, must be declared immediately post procedure. Clinical follow-up will be performed at 30 days.

Telephone follow-ups will be performed at 6 months and 1 year post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an indication for PCI including angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, or recent STEMI. For STEMI the time of presentation to the first treating hospital, whether a transfer facility or the study hospital, must be >24 hours prior to enrollment and enzyme levels (CK-MB or Troponin) demonstrating that either or both enzyme levels have peaked.
2. Non-target vessel PCI are allowed prior to enrollment depending on the time interval and conditions as follows:

   During Baseline Procedure:

   PCI of non-target vessels performed during the baseline procedure itself immediately prior to enrollment if successful and uncomplicated defined as: <50% visually estimated residual diameter stenosis, TIMI Grade 3 flow, no dissection ≥ NHLBI type C, no perforation, no persistent ST segment changes, no prolonged chest pain, no TIMI major or BARC type 3 bleeding.

   Less than 24 hours prior to Baseline Procedure:

   Not allowed (see exclusion criteria #2). 24 hours-30 days prior to Baseline Procedure: PCI of non-target vessels 24 hours to 30 days prior to enrollment if successful and uncomplicated as defined above.

   In addition, in cases where non-target lesion PCI has occurred 24-72 hours prior to the baseline procedure, at least 2 sets of cardiac biomarkers must be drawn at least 6 and 12 hours after the non-target vessel PCI.

   If cardiac biomarkers are initially elevated above the local laboratory upper limit of normal, serial measurements must demonstrate that the biomarkers are falling.

   Over 30 days prior to Baseline Procedure:

   a. PCI of non-target vessels performed greater than 30 days prior to procedure whether or not successful and uncomplicated.
3. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

   Angiographic inclusion criteria (visual estimate):
4. Target lesion(s) must be located in a native coronary artery or bypass graft conduit with visually estimated diameter of ≥2.5 mm to ≤4.25 mm.
5. Complex lesions are allowed including calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), presence of thrombus, CTO, bifurcation lesions (except as noted in exclusion criteria #30), ostial RCA lesions, tortuous lesions, bare metal stent restenotic lesions, protected left main lesions, and saphenous vein graft lesions.
6. Overlapping stents are allowed.

Exclusion Criteria:

General Exclusion Criteria:

1. STEMI within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital or in whom enzyme levels (either CK-MB or Troponin) have not peaked.
2. PCI within the 24 hours preceding the baseline procedure.
3. Non-target lesion PCI in the target vessel within 12 months of the baseline procedure.
4. History of stent thrombosis.
5. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
6. Subject is intubated.
7. Known LVEF <30%.
8. Relative or absolute contraindication to DAPT for 6 months in non-ACS patients and 12 months in ACS patients (including planned surgeries that cannot be delayed, or subject is indicated for chronic oral anticoagulant treatment).
9. Calculated creatinine clearance <30 mL/min using Cockcroft-Gault equation (<40 mL/min for subjects participating in the angiographic follow-up sub-study).
10. Hemoglobin <10 g/dL.
11. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
12. White blood cell (WBC) count <3,000 cells/mm3.
13. Clinically significant liver disease.
14. Active peptic ulcer or active bleeding from any site.
15. Bleeding from any site within the prior 8 weeks requiring active medical or surgical attention.
16. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.
17. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
18. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
19. Known allergy to the study stent components, cobalt, nickel, chromium, molybdenum, Carbosil®, PBMA, polymer, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
20. Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (clopidogrel, prasugrel, ticagrelor), or heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated.
21. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease).
22. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
23. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within one week before treatment).
24. Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
25. Patient has received an organ transplant or is on a waiting list for an organ transplant.
26. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.
27. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

    Angiographic Exclusion Criteria (visual estimate):
28. More than 100 mm length of planned stenting in the entire coronary tree.
29. Unprotected left main lesions ≥30%, or planned left main intervention.
30. Ostial LAD or LCX lesions (stenting of any diseased segment within 5 mm of the unprotected left main coronary artery).
31. Bifurcation lesions with planned dual stent implantation.
32. Stenting of lesions due to DES restenosis.
33. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the baseline procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abid Assali, Prof. MD, Principal Investigator — Rabin Medical Center; Shmuel Banai, Prof. MD, Principal Investigator — Souraski Medical Center; Michael Jonas, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BioNIR Drug Eluting Stent System
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BioNIR Drug Eluting Stent System
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Israel | 58

OUTCOME MEASURES:

1. Primary Outcome: Device Success in the Target Lesion as Determined by the Angiographic Core Laboratory
Time Frame: during baseline procedure
Measure: Count of Participants; unit: Participants
Arm/Group | BioNIR Drug Eluting Stent System
Number analyzed (Participants) | 58
Participants | 58

2. Secondary Outcome: Target Lesion Success
Description: Lesion success is defined as achievement of a final in-stent residual diameter stenosis of <50% (by QCA) using any percutaneous method.
Time Frame: during baseline procedure
Reporting Status: Not Posted

3. Secondary Outcome: Procedure Success
Description: Procedure success is defined as achievement of a final in-stent diameter stenosis of <50% (by QCA) using the assigned device and/or with any adjunctive devices, without the occurrence of cardiac death, Q wave or non-Q wave MI, or repeat revascularization of the target lesion during the hospital stay.
Time Frame: during baseline procedure
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Major Adverse Cardiac Events (MACE)
Time Frame: Clinical follow-up will be performed at 30 days.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Major Adverse Cardiac Events (MACE)
Time Frame: Telephone follow up will be performed at 6 months post procedure
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Major Adverse Cardiac Events (MACE)
Time Frame: Telephone follow up will be performed at 1 year post procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The Investigator monitored the occurrence of adverse events or device deficiencies for each subject during the whole course of the trial, baseline and post procedure, 30 days, 6 months and 1 year.
Arm/Group | BioNIR Drug Eluting Stent System
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 3/58
Other Adverse Events (participants affected / at risk) | 16/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BioNIR Drug Eluting Stent System (N=58)
Peri procedureal MI (Cardiac disorders) | 2
Non specific chest pain (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BioNIR Drug Eluting Stent System (N=58)
Viral Infection (Infections and infestations) | 1
General disorders and administration site conditions (General disorders) | 6
Cardiac disorders (Cardiac disorders) | 6
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2
eye disorders (Eye disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No